CLINICAL TRIAL: NCT02690077
Title: Family-Centered Cesarean: A Randomized Controlled Trial
Brief Title: Family-Centered Cesarean Delivery
Acronym: FCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 02-16
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Results first posted 2023-03-31 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-04

CONDITIONS: Patient Satisfaction; Earlier Family Bond Initiation; Maternal and Neonatal Outcomes
Keywords: Patient Satisfaction; Earlier Family Bond Initiation; Maternal and Neonatal Outcomes
MeSH Terms: conditions — Patient Satisfaction | interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Method 1 by Preference 1 (Active Comparator): Delivery through the Family-Centered Cesarean for patients with known Family-Centered preference.
  Interventions: Procedure: Family-Centered Cesarean
- Method 1 by Preference 2 (Active Comparator): Delivery through the Family-Centered Cesarean for patients with known Traditional Cesarean preference.
  Interventions: Procedure: Family-Centered Cesarean
- Method 2 by Preference 1 (Active Comparator): Delivery through the Traditional Cesarean for patients with known Family-Centered preference.
  Interventions: Procedure: Traditional Cesarean
- Method 2 by Preference 2 (Active Comparator): Delivery through the Traditional Cesarean for patients with known Traditional Cesarean preference.
  Interventions: Procedure: Traditional Cesarean

INTERVENTIONS:
Procedure: Family-Centered Cesarean — Procedure involves lowering part of the surgical drape exposing a transparent window through which the mother can watch the birth of her baby; the baby will be placed on her chest immediately after the delivery. Cleaning and evaluation of the baby will be done by a nurse who is standing at the head of the bed.
  Other Names: Gentle Cesarean
  Arms: Method 1 by Preference 1; Method 1 by Preference 2
Procedure: Traditional Cesarean — Procedure involves keeping the surgical drape up throughout the entire surgery so that the birthing process will not be visible to the mother, and the baby will be taken to the warmer to be evaluated and cleaned after birth but is available to be laid on the mother's chest at any point upon request.
  Other Names: Cesarean Section
  Arms: Method 2 by Preference 1; Method 2 by Preference 2

SUMMARY:
The purpose of this study is to determine if patient birthing experiences differ between the family-centered and traditional cesarean methods. We hypothesize that the family-centered cesarean method will lead to more unique and personalized cesarean birthing experiences without increasing the risks of adverse neonatal and maternal outcomes from those documented with the traditional cesarean.

DETAILED DESCRIPTION:
Patients will be consented and randomized to one of two delivery methods by the research coordinator, resident physician, charge nurse or nurse on the day of their planned cesarean section. Several variables of interest will be collected via the electronic medical record and within the OR. Additionally, assessment of patient satisfaction will be conducted following delivery. Questions from an 11-item questionnaire will be asked of the patient by the study coordinator, resident physician, nurse or charge nurses.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age
* Women with planned cesarean section
* ≥38 weeks of gestation
* Singleton fetus
* Reassuring fetal status (status of scheduled, green and some yellow

Exclusion Criteria:

* Women with an urgent or emergency clinical situation in which the medical staff caring for the patient determines that obtaining consent would interfere with the patient's clinical care
* Patients that decline to consent to participate (an opt out log including the consenters initials, time of day, and reason is kept)
* Patients with anticipated heavy intraoperative bleeding (bleeding disorders, placenta previa, suspected placenta abruption, etc.)
* Known maternal co-morbidities that could impact neonatal well-being (e.g., uncontrolled diabetes, etc.)
* Chorioamnionitis or prolonged rupture of membranes (≥18 hours in duration)
* Known fetal anomalies
* BMI ≥45 kg/m2
* Estimated fetal weight <2000 grams

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie M Forgie, DO, Principal Investigator — Aurora Health Care, Inc.
Locations (2):
- United States (2):
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armbrust R, Hinkson L, von Weizsacker K, Henrich W. The Charite cesarean birth: a family orientated approach of cesarean section. J Matern Fetal Neonatal Med. 2016;29(1):163-8. doi: 10.3109/14767058.2014.991917. Epub 2015 Jan 9. PMID 25572878
- [Background] Smith J, Plaat F, Fisk NM. The natural caesarean: a woman-centred technique. BJOG. 2008 Jul;115(8):1037-42; discussion 1042. doi: 10.1111/j.1471-0528.2008.01777.x. PMID 18651885
- [Background] Magee SR, Battle C, Morton J, Nothnagle M. Promotion of family-centered birth with gentle cesarean delivery. J Am Board Fam Med. 2014 Sep-Oct;27(5):690-3. doi: 10.3122/jabfm.2014.05.140014. PMID 25201938
- [Background] de Alba-Romero C, Camano-Gutierrez I, Lopez-Hernandez P, de Castro-Fernandez J, Barbero-Casado P, Salcedo-Vazquez ML, Sanchez-Lopez D, Cantero-Arribas P, Moral-Pumarega MT, Pallas-Alonso CR. Postcesarean Section Skin-to-Skin Contact of Mother and Child. J Hum Lact. 2014 Aug;30(3):283-286. doi: 10.1177/0890334414535506. Epub 2014 May 20. PMID 24847031
- [Background] Moran-Peters JA, Zauderer CR, Goldman S, Baierlein J, Smith AE. A quality improvement project focused on women's perceptions of skin-to-skin contact after cesarean birth. Nurs Womens Health. 2014 Aug-Sep;18(4):294-303. doi: 10.1111/1751-486X.12135. PMID 25145718
- [Result] Kram JJF, Montgomery MO, Moreno ACP, Romdenne TA, Forgie MM. Family-centered cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Nov;3(6):100472. doi: 10.1016/j.ajogmf.2021.100472. Epub 2021 Aug 26. PMID 34454161

RESULTS

PARTICIPANT FLOW:
Groups:
- Method 1 (Family-Centered Cesarean): Delivery through the Family-Centered Cesarean.
  Family-Centered Cesarean: Procedure involves lowering part of the surgical drape exposing a transparent window through which the mother can watch the birth of her baby; the baby will be placed on her chest immediately after the delivery. Cleaning and evaluation of the baby will be done by a nurse who is standing at the head of the bed.
- Method 2 (Traditional Cesarean): Delivery through the Traditional Cesarean.
  Traditional Cesarean: Procedure involves keeping the surgical drape up throughout the entire surgery so that the birthing process will not be visible to the mother, and the baby will be taken to the warmer to be evaluated and cleaned after birth but is available to be laid on the mother's chest at any point upon request.
Period: Overall Study
Arm/Group | Method 1 (Family-Centered Cesarean) | Method 2 (Traditional Cesarean)
Started | 73 | 76
Completed | 68 | 61
Not Completed | 5 | 15
Not completed — Excluded from analyses for no OR worksheet or questionnaire completed | 5 | 8
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Excluded by IRB | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Method 1 (Family Centered Cesarean): Delivery through the Family-Centered Cesarean.
  Family-Centered Cesarean: Procedure involves lowering part of the surgical drape exposing a transparent window through which the mother can watch the birth of her baby; the baby will be placed on her chest immediately after the delivery. Cleaning and evaluation of the baby will be done by a nurse who is standing at the head of the bed.
- Total: Total of all reporting groups
Arm/Group | Method 1 (Family Centered Cesarean) | Method 2 (Traditional Cesarean) | Total
Number analyzed (Participants) | 68 | 61 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.6) | 29.5 (5.2) | 29.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 61 | 129
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 26 | 20 | 46
  Black non-Hispanic | 27 | 24 | 51
  Hispanic | 12 | 15 | 27
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: 11-item Patient Satisfaction Questionnaire
Description: The primary objective of this study was to compare satisfaction with birthing experiences between women who underwent either a family-centered or traditional cesarean delivery, using a modified Likert scale, ranging from 1 (lowest) to 5 (highest).
Time Frame: Assessed at time of discharge from the hospital (typically 3-5 days post-delivery)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Method 1 (Family-Centered Cesarean) | Method 2 (Traditional Cesarean)
Number analyzed (Participants) | 68 | 61
units on a scale
  How satisfied were you with your involvement with the delivery of the baby? | 4.6 (0.8) | 4.4 (0.9)
  Did the method for delivery meet your expectations? | 4.6 (0.7) | 4.3 (1.0)
  Based on previous cesarean delivery how satisfied are you with the method of delivery of your baby? | 4.9 (0.7) | 4.7 (1.0)

2. Secondary Outcome: Timing of Initiation of Family Bond Following Delivery
Description: The secondary objective of this study is to determine if there is a difference in time-to-initiation of family bond between the family-centered cesarean delivery method and traditional cesarean delivery method.
Time Frame: Assessed in Operating Room
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Method 1 (Family-Centered Cesarean) | Method 2 (Traditional Cesarean)
Number analyzed (Participants) | 68 | 61
minutes | 5.1 (17.2) | 16.3 (13.9)

3. Secondary Outcome: Number (Percent) of Patients Planning to Breastfeeding After Discharge
Description: The tertiary objective of this study is to determine if breastfeeding was more likely to occur between the family-centered cesarean delivery method and traditional cesarean delivery method.
Time Frame: Assessed at time of discharge from the hospital (typically 3-5 days post-delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Method 1 (Family-Centered Cesarean) | Method 2 (Traditional Cesarean)
Number analyzed (Participants) | 68 | 61
Participants | 47 | 33

ADVERSE EVENTS:
Time Frame: 2 years, 1 month (participants were followed through discharge).
Description: No adverse events were noted.
Arm/Group | Method 1 (Family Centered Cesarean) | Method 2 (Traditional Cesarean)
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/76
Other Adverse Events (participants affected / at risk) | 0/73 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT02690077/Prot_SAP_000.pdf